CLINICAL TRIAL: NCT02860117
Title: The Effectiveness of Ketamine Continuous Infusion on Opioid Consumption and Pain Management in Severe Burned Patients, a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Ketamine Continuous Infusion on Opioid Consumption and Pain Management in Severe Burned Patients
Acronym: ccimb
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: change in hospital policy
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Felipe Chiodini Machado, Anesthesiologist, Member of USaoPauloGH Pain Management staff, Principal investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1551628
Record Dates: First submitted 2016-07-26; First posted 2016-08-09 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Pain, Burning
Keywords: ketamine; continuous infusion; severe burned patients
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketatamine (Active Comparator): Ketamine continuous infusion 0,2mg/kg/h
  Interventions: Device: Ketamine continuous infusion
- Placebo (Placebo Comparator): Placebo in continuous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Device: Ketamine continuous infusion — Ketamine 0.1% 250mL continuous infusion (0,2ml/kg/h)
  Other Names: Ketamine
  Arms: Ketatamine
Drug: Placebo — Placebo continuous infusion (0,2 ml/kg/h)
  Other Names: NaCl 0,9%
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of ketamine in continuous infusion in the control of pain intensity, the impact on the consumption of opioids and observe the side effect profile in patients suffering from great extent of burns.

DETAILED DESCRIPTION:
Despite advances in pharmacology and in analgesic techniques, pain in burned patients is unwieldy yet, this occurs in such cases due to the complexity and intensity and the need for multidisciplinary medical team. The burn pain is classified as nociceptive, but can also present a neuropathic component. Overall this is a pain at rest and during movement, being aggravated by procedures like changing dressings. In the weeks after the burn there is intense pain due to injury and the management of the framework, which often involves dressing changes and other procedures such as surgery in donor area skin.

The use of opioids in high doses can lead to unwanted side effects.To reduce the adverse effects resulting from the use of opioids in high doses, we purpose the use of intravenous continuous infusion of ketamine. In controlling the pain of major burned patient there is evidence only of the use of ketamine in the form of intermittent boluses, especially during dressing changes or in the perioperative period. The use of ketamine in continuous infusion lacks evidence in this group of patients The purpose of this study is to evaluate the efficacy of ketamine in continuous infusion in the control of pain intensity, the impact on the consumption of opioids and observe the side effect profile in patients suffering from great extent of burns.

ELIGIBILITY:
Inclusion criteria will be considered:

1. patients admitted to the burn unit of the Clinical Hospital with burnt body area of 25% or more;
2. aged between 18 and 60 years;
3. with surgical risk classification according to the "American Society of Anesthesiologists' (ASA) I and II;
4. has no known allergy or any other contraindications of the drugs that are used in the treatment protocol;
5. hemodynamically stable, considering systolic blood pressure greater than 90 mmHg;
6. with preserved consciousness level, measured by the Glasgow coma scale, with a score equal to 15;
7. with the possibility of drug administration orally or by naso-gastric tube

Exclusion criteria will be considered:

1. patients younger than 18 or older than 60 years;
2. with surgical risk classification according to the "American Society of Anesthesiologists' (ASA) III or higher;
3. with known allergy or any contraindications of the drugs that are used in the treatment protocol;
4. patients with q chronic pain or chronic analgesic users prior to burning in treatment;
5. hemodynamically unstable, considering systolic blood pressure below 90 mm Hg;
6. with changing level of consciousness;
7. without the possibility of administering drugs orally or by nasogastric tube.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | up to 10 days
  Rescue analgesic demand will be evaluated through patient controlled analgesia device up to 10 days of intervention

SECONDARY OUTCOMES:
Side effects questionnaire | up to 10 days
  the research team using a side effects questionnaire based on the major ketamine and opioid side effects

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Palmeira, MD, PhD, Study Director — University of Sao Paulo General Hospital
Locations (1):
- Hospital das Clínicas da FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No